CLINICAL TRIAL: NCT04100577
Title: Addressing Black Infant Mortality in Wisconsin Through a Collaborative Health Equity Approach Through Community Based Group Prenatal Care and Infant Support
Brief Title: Today Not Tomorrow Pregnancy and Infant Support Program (TNT- PISP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0684; A536784 (Other: UW Madison); SMPH\PEDIATRICS\NEWBORN NURS (Other: UW Madison); Protocol Version 3/5/2020 (Other: UW Madison)
Record Dates: First submitted 2019-09-19; First posted 2019-09-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Infant Mortality; Infant Death; Racial Bias; Prenatal Stress; Prenatal Care; Maternal Child Health; Health Problems in Pregnancy; Adverse Childhood Experiences; Mental Health; Support Groups; Minority Health; Healthcare Disparities; Maternal-child Health Services; Social Determinants of Health; Trust; Physician-Patient Relations; Quality of Care
Keywords: TNT-PISP
MeSH Terms: conditions — Infant Death; Racism; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A longitudinal, quasi-experimental design with two study arms will be used. Study arm 1 will consist of self-identified pregnant black women who are enrolled in the TNT-PISP intervention and Study arm 2 will consist of self-identified pregnant black women who are not enrolled in the TNT-PISP intervention. During the recruitment process, potential study participants will be able to self- select which study arm they would like to be in after each arm is described in detail. Although self-selection is traditionally discouraged in research, given the vulnerable population the investigator will be working with and historic distrust with medical community, investigator believe there is power in giving women of color choice in how they wish to navigate and engage with this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNT PISP intervention (Experimental): Participants in TNT PISP intervention group will come to once monthly educational support group sessions and will be additionally enrolled in the community based doula program where they will receive 1 on 1 doula and lactation support throughout their pregnancy, delivery, and postpartum period. They will receive prenatal care clinical visits on their own with their prenatal care provider. In phase 2 of the study, participants will be offered on site prenatal care once per month.
  Interventions: Other: Today Not Tomorrrow Pregnancy and Infant Support Program
- Control (No Intervention): Participants in control group will have no enhanced prenatal care support. They will attend visits on their own with their prenatal care provider and participation in this research study will not interfere with the prenatal care.

INTERVENTIONS:
Other: Today Not Tomorrrow Pregnancy and Infant Support Program — The Today Not Tomorrow Pregnancy and Infant Support Program (TNT-PISP) is a collaborative community-based support group uniquely designed to serve black women and infants through once monthly group sessions delivered prenatally and in the immediate postpartum period.
  Arms: TNT PISP intervention

SUMMARY:
This pilot project aims to implement and investigate the feasibility and acceptability of a unique community based prenatal care and support model for African American women and infants in Dane County. The model, the "Today Not Tomorrow Pregnancy and Infant Support Program (TNT-PISP)" builds on emerging evidence about how to effectively implement and sustain prenatal care in black communities. It combines three approaches-community-based doula programs; group-based models of prenatal care, such as Centering Pregnancy; and community-based pregnancy support groups-into once monthly group sessions held during the prenatal and immediate postpartum period. The project is based at the Today Not Tomorrow Family Resource Center in Madison's East Side Community Center, and carried out in close collaboration with Project Babies, Harambee Village Doulas, and the African American Breastfeeding Alliance of Dane County, Inc.

DETAILED DESCRIPTION:
Wisconsin leads the nation in the number of African American babies dying before their 1st birthday. These deaths are primarily due to complications of prematurity - babies being born too early and too soon. Additionally, Wisconsin's black infant mortality rate is significantly higher than that of whites and represents a serious health inequity that is critical for local research and advocacy efforts to address. The factors leading to inequities in preterm birth and infant mortality are complex and multifactorial; therefore, multidisciplinary and innovative approaches to prenatal and inter conception care are critical to improve these outcomes.

Previous research and feedback from black women living in Dane County has shown that lack of social support and culturally relevant models of preconception, prenatal, and inter-conception care has been a barrier to optimal quality of care and maternal child health outcomes. Further research has demonstrated that evidence based intervention approaches used nationally such as a) community-based doula programs, b) group-based models of prenatal care such as Centering Pregnancy, and c) community-based pregnancy and inter conception support groups hold promise as relevant prevention strategies, yet there are many barriers to their effective adoption in communities of color.

In response to the current birth outcome inequities that exist in Wisconsin, the objective of the current proposal is to implement and investigate a novel approach that combines aspects of all three of the above-mentioned evidence-based models and builds upon emerging evidence about how to effectively implement and sustain prenatal care interventions in Black communities: the TNT-PISP. The TNT-PISP approach is based on increasing evidence that models of prenatal care that are community driven, group based, culturally relevant, family centered, and include enhanced social support have the potential to significantly decrease African American prematurity rates and improve other maternal and infant health measures.

TNT-PISP is a collaborative community-based support group uniquely designed to serve black women and infants through once monthly group sessions delivered prenatally and in the immediate postpartum period. Each 2 hour TNT-PISP session will be held at the Today Not Tomorrow Family Resource Center located on Madison's Eastside and will be led by local African American community-based doulas supported by and in collaboration with a host of other community partners and healthcare professionals from diverse backgrounds. Each session will consist of food, hands on learning activities, peer to peer socio-emotional support, guest speakers, relationship building activities, and dynamic discussions on a host of pregnancy and newborn care related topics. In addition to group sessions, participants will be additionally have the option to be enrolled in a community based doula program to receive support outside the group sessions, and culturally sensitive mental health and case management support services on an as-needed basis. Via partnerships with various healthcare providers and systems, there are also tentative plans for future expansion so that select participants will additionally be able to receive their prenatal care exams on site.

Assessments with individual participants in each study arm will occur at three contact points: At start of pregnancy, around time of birth/early postpartum and ~ 6 months postpartum. At each time of contact, they will be asked to complete a series of questionnaires and participate in a semi-structured interview with PI. If additionally consented, medical records of all study participants will be analyzed to assess secondary outcomes.

This is a pilot study. As the study transition to larger scale efficacy trials in future, it will be important to be able to link to and review patient perinatal outcomes. Feasibility questions asked in this study are 1) Will it be obvious who meets and who does not meet our eligibility criteria? Are the eligibility criteria sufficient or too restrictive? 2) Will our study questionnaires and data collection tools be easy to understand and user friendly? 3) What systems levels facilitators and barriers will contribute to the implementation and success of this pilot program? 4) Will participants be pleased with the curriculum/design of the TNT-PISP pilot intervention? Is delivering prenatal care on site something participants would find beneficial in addition to group education/support sessions? 5) Will our team have the capacity to implement and maintain the TNT-PISP program? Part of the feasibility trial of this study is assessing how receptive mothers are to us accessing their medical records and data retrieval logistics. Additionally, semi structured interviews with up to 10 key academic/community based stakeholders involved in the implementation process of TNT-PISP program will be obtained and evaluated via thematic analysis. Interviews with these key stakeholders will not be compensated and will be on a volunteer basis. These interviews will collect information on the facilitators and barriers to implementing and maintaining the program from their standpoint.

Finally, two focus groups will occur over the course of the study period. The first focus group will involve self-identified black women living in Dane County interested in providing feedback on the ideal design of a culturally relevant community based prenatal care and support program such as the TNT-PISP pilot. The second focus group will be limited to research participants who participated in the TNT PISP intervention for at least 1 session and will provide feedback on facilitators and barriers to its acceptability and feasibility as well as preliminary feedback on maternal child health outcomes and attitudes impacted as a result of the program. All individuals involved in conducting one on one interviews/focus groups will be women of color on the research team to facilitate comfort and trust for the participants.

All focus groups and individual interviews will be audio recorded.

One on one interviews will occur either on the phone or at a comfortable public location of the subject's desire (ex: library or at the TNT Family Resource Center). One on one interviews will take place in a private room to ensure as much privacy as possible. Subjects will also have the option for the interview to occur in their home and if that occurs, they will be made aware that the interviewer is a mandatory reporter if any concerning activities in the home were to be observed.

The focus groups will take place at the TNT-Family Resource Center. All one on one interviews will be conducted by Dr. Zapata. All focus groups will be conducted by Dr. Zapata in collaboration with other research team members listed in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant self- identified black women
* Living in Dane County Wisconsin

Exclusion Criteria:

* Not pregnant or did not deliver within the last year
* Do not self- identify as a black woman

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Participant recruitment as assessed by percentage of participants enrolled in Today Not Tomorrow Pregnancy and Infant Support Program (TNT-PISP) | 2 years
  TNT-PISP is aiming to recruit 20 self-identified African American women into the TNT-PISP Pilot. The actual recruitment will be measured as percentage of participants recruited, assuming recruitment of 20 participants per arm as 100%
Retention rate of participants as assessed by percentage of participants adhered to study for 2 years | 2 years
  Retention rate of participants as assessed by percentage of participants adhered to study for 2 years

SECONDARY OUTCOMES:
Preliminary Maternal Child Health Outcomes: Birth weight | At child birth or at 38 week average gestation time whichever will come first
  Birth weight of baby will be assessed from the medical records in the TNT-PISP group and the control group to assess the effect of the intervention on the preliminary maternal child health outcome.
Preliminary Maternal Child Health Outcomes: Birth gestational age | At child birth or at 38 week average gestation time whichever will come first
  Birth gestational age will be assessed from the medical records in the TNT-PISP group and the control group to assess the effect of the intervention on the preliminary maternal child health outcome.
Percentage of participants breastfed babies at time of birth | up to 2 years
  Percentage of participants breastfed babies at time of birth as per the medical records
Percentage of participants opted for inter-conception care plans | 2 years
  Percentage of participants opted for inter-conception care plans as per the medical records
Rate of attendance to 6- week postpartum visit | 6 week postpartam
  Rate of attendance to 6- week postpartum visit as per the medical records

CONTACTS AND LOCATIONS:
Overall Officials: Jasmine Y Zapata, MD, MPH, Principal Investigator — University of WI School of Medicine and Public Health
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No